CLINICAL TRIAL: NCT00536848
Title: The Effect of Probiotic Supplementation With Lactobacillus GR-1 and RC-14,on the Immune Status, Diarrhea and Bacterial Vaginosis Cure Rate Among HIV Patients; a Randomised, Placebo Controlled Trial
Brief Title: The Effect of Probiotics on the Immune Status, Diarrhea and Bacterial Vaginosis Cure Rate Among HIV Patients
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Institute for Medical Research, Tanzania (Other Government)
Collaborators: University of Western Ontario, Canada (Other); Erasmus Medical Center (Other); Sekou-Toure Regional Hosipital, Mwanza, Tanzania (Unknown); London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other); Danone Institute International (Other)
Responsible Party: Director, National Institute for Medical Research, Mwanza research centre
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MRRC HIV-Probiotics15
Record Dates: First submitted 2007-09-27; First posted 2007-09-28 (Estimated); Last update posted 2009-01-30 (Estimated); Status verified 2009-01

CONDITIONS: HIV Infections; Diarrhea; Bacterial Vaginosis
Keywords: Probiotics; HIV; AIDS; Diarrhea; Lactobacillus rhamnosus GR-1; Lactobacillus reuteri RC-14; Immune system; Infectious Diseases; Complementary Therapies; Treatment Naive
MeSH Terms: conditions — HIV Infections; Diarrhea; Vaginosis, Bacterial; Acquired Immunodeficiency Syndrome; Communicable Diseases | interventions — Metronidazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): Metronidazole for 10 days, probiotics for 6 months
  Interventions: Dietary Supplement: Lactobacillus rhamnosus GR-1 + Lactobacillus reuteri RC-14; Drug: Metronidazole
- B (Placebo Comparator): Metronidazole for 10 days, placebo for 6 months
  Interventions: Dietary Supplement: Placebo; Drug: Metronidazole

INTERVENTIONS:
Dietary Supplement: Lactobacillus rhamnosus GR-1 + Lactobacillus reuteri RC-14
  Arms: A
Dietary Supplement: Placebo
  Arms: B
Drug: Metronidazole

SUMMARY:
The purpose of this study is to asses whether probiotics Lactobacillus rhamnosus (GR-1) and reuteri (RC-14) are able to prevent diarrhea, delay the decline of the immune system and prevent and/or cure bacterial vaginosis among HIV patients.

DETAILED DESCRIPTION:
Background: Two third of all people infected with HIV live in Sub-Saharan Africa. A region also affected with a great burden of other infectious diseases. Relatively few patients have access to anti-retroviral treatment and many suffer from debilitating diarrhea that causes their immune system to deteriorate. Prevention of infectious diseases among HIV patients is of great importance and makes the immune system deteriorate less rapidly. The track record for probiotics to prevent and alleviate infectious diarrhea is impressive. So, the use of probiotics among HIV patients is a logical step and could be an adjunctive tool for physicians to halt the decline of the CD4 count.

Another important application for the use of probiotics is in the treatment of bacterial vaginosis (BV). BV is a vaginal infection, caused by a group of pathogens, which is extremely common, and estimated to occur in 50% of black African women. In the US, the prevalence is 29%, which again is extremely high. This infection makes a woman more vulnerable to contracting sexually transmitted infections, including HIV. Having BV is also a risk factor to transmit HIV to a partner or a newborn. Conventional antibiotic treatment of BV has a cure rate of 40% among black African women. A recent study shows that combining the probiotic strains Lactobacillus rhamnosus GR-1 and Lactobacillus reuteri RC-14 with an antibiotic has a cure rate of 88%.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed HIV infection.
* Participant does not meet the criteria for ARV therapy, CD4 count > 200, no clinical stage 3 or 4 [National guidelines, 2005].
* Having an intermediate Nugent score (4-6), or a positive Nugent score (7-10).

Exclusion Criteria:

* Pregnancy or lactating.
* Menstruation at time of diagnosis.
* Hypersensitive to metronidazole/warfarin/lithium/disulfiram.
* Not willing to avoid alcohol use during the metronidazole treatment of 10 days.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 65 (Actual)
Dates: Start 2007-10; Primary Completion 2008-08 (Estimated); Study Completion 2008-08 (Estimated)

PRIMARY OUTCOMES:
CD4 count | assessed at 10 and 25 weeks

SECONDARY OUTCOMES:
Bacterial vaginosis cure rate | assesed at week 2, 5, 15, 25
Total serum IgE levels | baseline and at 10 weeks
Serum cytokine levels | baseline and at 10 weeks
Diarrhea incidence and length of episodes | 25 weeks

CONTACTS AND LOCATIONS:
Overall Officials: John Changalucha, MSc, Principal Investigator — National Institute for Medical Research, Mwanza Research Centre
Locations (1):
- Sekou-Toure Regional Hospital, Mwanza, Tanzania

REFERENCES:
- [Derived] Hummelen R, Changalucha J, Butamanya NL, Cook A, Habbema JD, Reid G. Lactobacillus rhamnosus GR-1 and L. reuteri RC-14 to prevent or cure bacterial vaginosis among women with HIV. Int J Gynaecol Obstet. 2010 Dec;111(3):245-8. doi: 10.1016/j.ijgo.2010.07.008. PMID 20801446
- See also: a project of the University of Western Ontario to bring probiotics to the developing world — http://www.westernheadseast.ca